CLINICAL TRIAL: NCT02587832
Title: Randomized Control Trial: Heated Humidity High Flow Nasal Cannula in Comparison With Nasal Continuous Positive Airway Pressure in the Management of Respiratory Distress Syndrome in Extreme Low Birth Infants in Immediate Post Extubation Period
Brief Title: High Flow Nasal Cannula in Comparison With Nasal Continuous Positive Airway Pressure in the Management of Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidra Medicine (Other)
Collaborators: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Mohammed Elkhwad, Principal investigator, Akron Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 081110
Record Dates: First submitted 2015-10-20; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Respiratory Distress Syndrome
Keywords: cpap; HHHFNC; RDS; ELBW
MeSH Terms: conditions — Respiratory Distress Syndrome; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HHHFNC (Active Comparator): Randomized to HHHFNC
  Interventions: Device: HHHFNC
- NCPAP (Active Comparator): Randomized to NCPAP
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: HHHFNC — Tri-Anim Vaptherm the Precision Flow, which is a self contained unit that provides flow rates up to or 8 LPM (Infants) of blended oxygen that is heated and humidified
  Other Names: VAPOTHERM
  Arms: HHHFNC
Device: NCPAP — Bubble CPAP System.
  Arms: NCPAP

SUMMARY:
To compare the primary outcome, failure of extubation defined by the need for re-intubation and mechanical ventilation within 5 days of initial extubation and secondary outcomes, morbidities and mortality after using of heated humidity high flow nasal cannula (HHHFNC) and Nasal Continuous Positive Airway Pressure (NCPAP) in the immediate post-extubation period for preterm infants between 24 and 28 weeks gestation with respiratory distress syndrome.

DETAILED DESCRIPTION:
Inclusion criteria were: 1) Preterm neonates with gestational age of 24 to 28 completed weeks. 2) In the case of twins, both neonates were included in the same treatment arm. 3) Success to wean with 24 hours to extubate. 4) Parental written informed consent for participation in the study obtained on admission into the hospital or prior to delivery.

Exclusion criteria were: 1) Evidence of severe birth asphyxia. 2) Known genetic or chromosomal disorders. 3) Infants delivered to mothers with ruptured membranes of more than three weeks duration. 4) Potentially life-threatening conditions unrelated to prematurity. 5) Participation in another clinical trial of any placebo, drug, biological, or device conducted under the provisions of a protocol.

Randomization A computer-generated block-randomization sequence with random block sizes was used. Infants who were part of multiple births underwent individual randomization. Clinicians opened consecutively numbered, sealed, brown envelopes immediately before extubation to determine the study-group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates with gestational age of 24 to 28 completed weeks.
2. In the case of twins, both neonates were included in the same treatment arm.
3. Success to wean with 24 hours to extubate.
4. Parental written informed consent for participation in the study obtained on admission into the hospital or prior to delivery.

Exclusion Criteria:

1. Evidence of severe birth asphyxia.
2. Known genetic or chromosomal disorders.
3. Infants delivered to mothers with ruptured membranes of more than three weeks duration.
4. Potentially life-threatening conditions unrelated to prematurity.
5. Participation in another clinical trial of any placebo, drug, biological, or device conducted under the provisions of a protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the need for re-intubation | 5 DAYS
  The primary outcome measured was failed extubation defined by the need for re-intubation and mechanical ventilation within five days of initial extubation.

SECONDARY OUTCOMES:
Duration of respiratory support using HHHFNC /NCPAP. | through study completion, an average of 1 year.
Incidence of nasal breakdown | through study completion, an average of 24 weeks
sepsis | through study completion, an average of 1 year.
intraventricular hemorrhage (IVH), | through study completion, an average of 24 weeks
retinopathy of prematurity (ROP) | through study completion, an average of 24 weeks
  number of participants with sepsis will be compared between the two arms. Sepsis was defined as a positive culture result from blood with concomitant clinical symptoms. Positive cultures were defined as having positive growth from the cerebrospinal fluid, tracheal, blood, or urine specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Elkhwad, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States